CLINICAL TRIAL: NCT07228117
Title: GATEWAY: Safety Evaluation of the MiniMed™ NMX8-AID System in Children and Adults Living With Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIP351
Record Dates: First submitted 2025-11-11; First posted 2025-11-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Arm 1 - No meal bolus administration (Experimental): Patients will be asked not to bolus for any of their meals while using the NMX8 pump.
  Interventions: Device: MiniMed™ NMX8-AID System with DS5™
- Arm 2 - Meal bolus administration at all meals (Experimental): Patients will be asked to bolus for all of their meals while using the NMX8 pump.
  Interventions: Device: MiniMed™ NMX8-AID System with DS5™
- Arm 3 - Meal bolus administration at will (Experimental): Patients are free to bolus or not bolus for their meals as they wish using NMX8 pump.
  Interventions: Device: MiniMed™ NMX8-AID System with DS5™

INTERVENTIONS:
Device: MiniMed™ NMX8-AID System with DS5™ — Patients will be provided with the NMX8 system with DS5 CGM.

SUMMARY:
The purpose of this study is to check that a new insulin pump, called NMX8, is safe when used with a continuous glucose monitoring sensor called Disposable Sensor 5 in people with diabetes. The study will include people with Type 1 diabetes who are 7-85 years old and people with Type 2 diabetes who are 18-85 years old. Patients will use their current therapy while also wearing the DS5 for up to 40 days. During this time, they will complete a meal and exercise log. Patients will then be put into one of three groups by a computer by chance and given the NMX8 pump to use for 90 days. During this time, patients will either bolus or not bolus for meals and continue to complete a meal and exercise log depending on the group they are in. Once their part in the study is over, if patients like the pump and want to keep using it, they may be able to join a Continued Access Period to keep using the NMX8 pump.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of screening according to diabetes type:

   1. T1D: Age 7-85 years
   2. T2D: Age 18-85 years
2. Has a clinical diagnosis of diabetes for a minimum per diabetes type below:

   1. T1D (Age 7-85 years): Diagnosis of T1D for at least 6 months, as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
   2. T2D (Age 18-85 years): Diagnosis of insulin-requiring T2D for 1 year or more, as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Is willing to provide informed consent/assent for participation.
4. Subject or parent/caregiver is literate and able to read the language (English or Spanish) offered in the study pump or study pump materials.
5. Is willing to wear the system continuously throughout the study.
6. Has a retinal eye examination prior to enrollment (if needed) per guidelines by the local professional society/hospital guidelines according to age, duration of diabetes and type of diabetes. Entry into the study is permitted at the investigators' discretion, depending on their interpretation of the findings.
7. Is willing to upload study pump data via an app or computer.
8. Is willing to take one of the following insulins and can financially support the use of insulin preparations as required by the study:

   1. Humalog™* (insulin lispro injection)
   2. NovoLog™*/NovoRapid™* (insulin aspart solution for injection)
   3. Admelog™* (insulin lispro injection)
   4. Merilog™* (insulin aspart)
   5. Authorized generic insulin aspart
   6. Authorized generic insulin lispro

Exclusion Criteria:

1. Unable to consent due to a mental or intellectual disability.
2. Has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following, during the 6 months prior to screening:

   1. Medical assistance (i.e., Paramedics, Emergency Room [ER] or Hospitalization)
   2. Coma or
   3. Seizures
3. Has a history of 1 or more episodes of diabetic ketoacidosis (DKA) in the last 6 months prior to screening visit.
4. T2D: Has had hyperglycemic hyperosmolar syndrome (HHS) in the last 6 months prior to screening visit.
5. Has any unresolved adverse skin condition in the area of sensor or infusion set placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
6. Currently pregnant or planning to become pregnant during the time period of study participation

   1. A negative pregnancy test will be required for all females of child-bearing potential prior to enrollment
   2. For sexually active females of child-bearing potential the investigator will use discretion to determine if the form of contraception that is being used is reliable
7. At investigator discretion, has hypothyroidism or hyperthyroidism that is not adequately treated.
8. Has diagnosis of adrenal insufficiency.
9. Has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit.
10. T1D: Is using non-insulin anti-hyperglycemic medication, other than metformin and/or Glucagon-like peptide-1 (GLP-1), in the 8 weeks prior to screening.

    1. Participants who have stopped using metformin and/or GLP-1 have done so at least 6 weeks prior to screening.
    2. Participants currently taking metformin and/or GLP-1 must be on a steady dose and remain on the same dose during study participation. Dose changes and reasons for changes will be documented throughout the study.
11. T2D: Is using non-insulin anti-hyperglycemic medication, other than metformin, GLP-1, Sodium-Glucose Cotransporter 2 (SGLT2) inhibitors, in the 8 weeks prior to screening.

    1. Participants who have stopped using metformin, GLP-1 or SLT-2 have done so at least 6 weeks prior to screening.
    2. Participants currently taking metformin, GLP-1 or SGLT-2 must be on a steady dose and remain on the same dose during study participation. Dose changes and reasons for changes will be documented throughout the study
12. Is using sulfonylureas and meglitinides, e.g. repaglinide
13. Is using inhalable insulin in the 8 weeks prior to screening.
14. Is using hydroxyurea at time of screening or plans to use it during the study
15. Is participating in another pharmaceutical or device trial within 2 weeks of enrollment or anticipates participation in another trial during the course of the study.
16. Is, at the discretion of the investigator, abusing drugs or alcohol.
17. Is, in the opinion of the investigator, not able to perform all study procedures safely.
18. Has a history of visual impairment which would not allow subject, even with the help of a caregiver, to participate in the study and perform all study procedures safely, as determined by the investigator.
19. Has elective surgery planned that requires general anesthesia during the course of the study.
20. Has sickle cell disease or other hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening.
21. Plans to receive red blood cell transfusion or erythropoietin over the course of study participation.
22. Is diagnosed with current eating disorder such as anorexia or bulimia.
23. Blood disorder or dyscrasia within 3 months prior to screening, which in the investigator's opinion could interfere with determination of HbA1c
24. Is on dialysis.
25. Has an estimated Glomerular Filtration Rate (eGFR) <30.
26. Has celiac disease that is not adequately treated as determined by the investigator.
27. Has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances.
28. Has had any of the following cardiovascular events more than 1 year prior to screening and should not participate at the discretion of the investigator: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances.
29. Is a member of the research staff involved with the study.
30. Is a Medtronic Diabetes employee or their immediate family member (excluding adult children and/or adult siblings).

Ages: 7 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall: Percent of Time in Range (TIR 70-180 mg/dL) | Throughout the study period, approximately 90 days.
  Percent of time in range (TIR 70-180 mg/dL) among all randomized subjects. Descriptive only.
Overall: Percent of Time in Hypoglycemia (< 70 mg/dL) | Throughout the study period, approximately 90 days.
  Percent of time in hypoglycemia (< 70 mg/dL) among all randomized subjects. Descriptive only.
Study Arm 1: Percent of Time in Range (TIR 70-180 mg/dL) | Throughout the study period, approximately 90 days.
  Percent of time in range (TIR 70-180 mg/dL) among subjects randomized to Study Arm 1. Descriptive only.
Study Arm 1: Percent of Time in Hypoglycemia (< 70 mg/dL) | Throughout the study period, approximately 90 days.
  Percent of time in hypoglycemia (< 70 mg/dL) among subjects randomized to Study Arm 1. Descriptive only.
Study Arm 2: Percent of Time in Range (TIR 70-180 mg/dL) | Throughout the study period, approximately 90 days.
  Percent of time in range (TIR 70-180 mg/dL) among subjects randomized to Study Arm 2. Descriptive only.
Study Arm 2: Percent of Time in Hypoglycemia (< 70 mg/dL) | Throughout the study period, approximately 90 days.
  Percent of time in hypoglycemia (< 70 mg/dL) among subjects randomized to Study Arm 2. Descriptive only.
Study Arm 3: Percent of Time in Range (TIR 70-180 mg/dL) | Throughout the study period, approximately 90 days.
  Percent of time in range (TIR 70-180 mg/dL) among subjects randomized to Study Arm 3. Descriptive only.
Study Arm 3: Percent of Time in Hypoglycemia (< 70 mg/dL) | Throughout the study period, approximately 90 days.
  Percent of time in hypoglycemia (< 70 mg/dL) among subjects randomized to Study Arm 3. Descriptive only.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (28):
  - Medical Investigations, Little Rock, Arkansas
  - Headlands Research California, LLC, Escondido, California
  - Sansum Diabetes Research Institute, Goleta, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco UCSF The Madison Clinic for Pediatric Diabetes, San Francisco, California
  - Mills-Peninsula Medical Center: Diabetes Research Institute, San Mateo, California
  - Stanford University Medical Center, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - USF Diabetes and Endocrinology Center, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Indiana University Health Riley Hospital for Children, Indianapolis, Indiana
  - Iowa Diabetes and Endocrinology Center, West Des Moines, Iowa
  - International Diabetes Center, Minneapolis, Minnesota
  - Bryan Physician Network, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYC Research Inc, Long Island City, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Revival Research Institute, Denton, Texas
  - Tekton Research, McKinney, Texas
  - Rainier Clinical Research Center, Renton, Washington
  - Seattle Children's, Seattle, Washington
- Australia (3):
  - John Hunter Children's Hospital, New Lambton, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - The Kids Research Institute Australia, Perth, Western Australia
- University of Otago - Dunedin Hospital, Dunedin, New Zealand

IPD SHARING:
Plan to Share IPD: No